CLINICAL TRIAL: NCT02782481
Title: A Multicenter, Randomized, Double-blind, Placebo Controlled, Parallel Group Clinical Study Investigating the Efficacy, Tolerability, and Safety of Continuous Subcutaneous ND0612 Infusion Given as Adjunct Treatment to Oral Levodopa in Patients With Parkinson's Disease With Motor Fluctuations
Brief Title: A Clinical Study Investigating the Efficacy, Tolerability, and Safety of Continuous Subcutaneous ND0612 Infusion Given as Adjunct Treatment to Oral Levodopa in Patients With Parkinson's Disease With Motor Fluctuations
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Decision to change the study design
Sponsor: NeuroDerm Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ND0612L-007
Record Dates: First submitted 2016-05-22; First posted 2016-05-25 (Estimated); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Levodopa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ND0612 High dose (Levodopa/Carbidopa solution) (Experimental): High dose ND0612 SC infusion over 24 h
  Interventions: Drug: ND0612
- ND0612 Low dose (Levodopa/Carbidopa solution) (Experimental): Low dose ND0612 SC infusion over 24 h
  Interventions: Drug: ND0612
- Placebo (Placebo Comparator): Placebo SC infusion over 24 h
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ND0612
  Other Names: Levodopa/Carbidopa solution
  Arms: ND0612 High dose (Levodopa/Carbidopa solution); ND0612 Low dose (Levodopa/Carbidopa solution)
Drug: Placebo
  Other Names: Placebo solution
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double blind, placebo controlled parallel group clinical study. Following a screening period of up to 28 days, eligible subjects will be randomized to receive adjunct treatment to oral LD/DDI (Dopa Decarboxylase Inhibitor) with continuous subcutaneous infusion of ND0612 or matching placebo for 16 weeks.

DETAILED DESCRIPTION:
This phase III randomized, double-blind, placebo controlled, parallel group clinical study will be conducted in 150 subjects with idiopathic PD who are experiencing motor complications despite optimized anti-PD therapy.

The study will investigate the efficacy, safety and tolerability of continuous SC infusion (16 weeks) of ND0612 compared with placebo infusion. The treatment period will be comprised of a 4-week adjustment period during which time the ND0612 infusion dose will remain constant and the oral LD/DDI dose can be decreased or increased back up to the Baseline levels. All other anti-PD treatments must remain constant. During the maintenance period (Weeks 5 to 16) all anti-PD medication including the ND0612/placebo should remain constant.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male and female PD subjects of any race aged 30-80 years
2. PD diagnosis consistent with the UK Brain Bank Criteria.
3. Modified Hoehn & Yahr scale in "ON" state ≤3
4. Subjects must experience motor fluctuations and experience an average of at least 2 hours daily in the "OFF" state
5. Taking at least 4 doses/day of IR LD/DDI (or at least 3 doses/day of Rytary) and taking, or having taken therapeutic doses of at least 2 other classes of anti-PD medications.
6. Subjects must be on stable doses of all their anti-PD medications for at least 28 days before Baseline (Day 1).
7. Subject and/or study partner must demonstrate ability to keep accurate diary entries of PD symptoms ("ON-OFF" diaries) with at least 75% concordance with the study rater by the end of the diary training session at the end of the screening period.
8. Mini Mental State Examination (MMSE) score >26.
9. Female subjects must be surgically sterile (hysterectomy, bilateral oophorectomy, or tubal ligation), postmenopausal (defined as cessation of menses for at least 1 year), or willing to practice a highly effective method of contraception.

Key Exclusion Criteria:

1. Atypical or secondary parkinsonism.
2. Psychosis or hallucinations in past 6 months.
3. Subjects with a clinically significant or unstable medical, surgical, psychiatric condition or laboratory abnormalities which, in the opinion of the Investigator or the EAC, represents a safety risk, makes the subject unsuitable for study entry or potentially unable to complete all aspects of the study.
4. Clinically significant ECG abnormalities.
5. Renal or liver dysfunction that may alter drug metabolism including Screening visit serum levels of creatinine >1.3 mg/dL, aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2x upper limit of normal (ULN), total bilirubin >2.5 mg/dL.
6. Positive serum serology for Hepatitits B Virus (HBV), Hepatitits C Virus (HCV) or Human Immunodeficiency Virus (HIV) at the Screening visit
7. Any malignancy in the 5 years prior to randomization excluding basal cell carcinoma of the skin or cervical carcinoma in situ that have been successfully treated
8. Use of prohibited medications as per protocol
9. Subjects who have previously undergone treatment for PD with a neurosurgical intervention (e.g., pallidotomy, thalamotomy, transplantation, deep brain stimulation procedures), Duodopa/Duopa, or continuous dopaminergic or apomorphine infusion.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
The change from Baseline to Week 16 in the mean percentage of "OFF" time during waking hours, based on patient's home diary assessments | baseline to week 16

CONTACTS AND LOCATIONS:
Locations (1):
- Haddasah Ein Kerem Medical center, Jerusalem, Israel